CLINICAL TRIAL: NCT07367906
Title: Effect of Digital Microlearning on Patient Safety Awareness and Clinical Decision-Making Among Nursing Students Before Surgical Clinical Practice: A Randomized Controlled Trial
Brief Title: Digital Microlearning and Patient Safety in Nursing Students
Acronym: DigiM-2026
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Volkan Gokmen, Assistant Professor, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Digital Microlearning-2026
Record Dates: First submitted 2026-01-13; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Medical Education; Patient Safety
Keywords: Digital microlearning; Nursing students; Patient safety awareness; Clinical error recognition; Surgical clinical practice; Educational intervention

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either a digital microlearning intervention group or a standard education control group and followed in parallel.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Microlearning Intervention Group (Experimental): Participants in this group will receive a patient safety-focused digital microlearning program before starting surgical clinical practice.
  Interventions: Behavioral: Digital Microlearning Program on Patient Safety
- Control Group Standard Education (No Intervention): Participants in this group will receive standard patient safety education as part of the undergraduate nursing curriculum without additional intervention.

INTERVENTIONS:
Behavioral: Digital Microlearning Program on Patient Safety — A structured digital microlearning program consisting of short, scenario-based modules (3-5 minutes each) focusing on patient safety awareness, clinical error recognition, prioritization, and clinical decision-making. The program will be delivered online for seven consecutive days before surgical clinical practice.
  Arms: Digital Microlearning Intervention Group

SUMMARY:
This randomized controlled study aims to evaluate the effect of a patient safety-focused digital microlearning program on nursing students before they begin surgical clinical practice.

Nursing students often face challenges related to patient safety and clinical decision-making during the transition from classroom learning to clinical settings. This study will examine whether short, structured digital learning modules can improve patient safety awareness, recognition of clinical errors, and decision-making skills.

Second-year undergraduate nursing students will be randomly assigned to either a digital microlearning intervention group or a control group receiving standard education. Outcomes will be measured before the intervention, immediately after the intervention, and during the first week of clinical practice.

DETAILED DESCRIPTION:
The transition from preclinical education to clinical practice represents a critical period for patient safety among nursing students. During this phase, limited clinical experience combined with increased responsibility may increase the risk of errors related to patient safety and clinical decision-making. Educational strategies that strengthen patient safety awareness and cognitive readiness before clinical exposure are therefore essential.

This study is designed as a single-center, parallel-group, randomized controlled trial. It will be conducted at the Faculty of Health Sciences, Department of Nursing, Agri Ibrahim Cecen University. Participants will consist of second-year undergraduate nursing students who are preparing to begin surgical clinical practice for the first time.

After baseline assessment, eligible participants will be randomly assigned to either an intervention group or a control group using stratified randomization based on gender and grade point average. The intervention group will receive a patient safety-focused digital microlearning program delivered online for seven consecutive days. The program consists of short, scenario-based modules lasting approximately 3-5 minutes each and addresses topics such as patient safety risks, clinical error recognition, prioritization, and decision-making under stress. Participants will be able to access the modules flexibly within a daily time limit.

The control group will receive standard patient safety education as part of the undergraduate nursing curriculum without additional intervention.

Outcome measures will be collected at three time points: baseline prior to the intervention (T0), immediately after completion of the intervention (T1), and during the first week of surgical clinical practice (T2). Primary outcomes include changes in patient safety awareness and clinical error recognition performance. Secondary outcomes include clinical decision-making under stress, perceived readiness for clinical practice, self-confidence, and acceptability of the digital microlearning program.

This study involves an educational intervention only and does not include any invasive procedures, drugs, or medical devices. Participation is voluntary, and written informed consent will be obtained from all participants. The study has been submitted for ethical review and will be conducted in accordance with ethical principles for research involving human participants.

ELIGIBILITY:
Inclusion Criteria:

* Second-year undergraduate nursing students
* Enrolled in the Faculty of Health Sciences, Department of Nursing
* Preparing to begin surgical clinical practice for the first time
* Aged 18 years or older
* Willing to participate and able to provide written informed consent

Exclusion Criteria:

* Previous surgical clinical practice experience
* Previous professional nursing or healthcare work experience
* Incomplete baseline assessment
* Declining to participate or withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient Safety Awareness | Baseline (T0): Prior to the educational intervention (Day 0) Post-intervention (T1): Within 1 week after completion of the intervention Follow-up (T2): During the first week of surgical clinical practice
  Change in patient safety awareness assessed using the Patient Safety Awareness Questionnaire, which evaluates students' understanding of patient safety principles, risk recognition, and safe clinical practices in surgical care. Outcome Measure: Total score on the Patient Safety Awareness Questionnaire, ranging from 0 to 100, where higher scores indicate greater patient safety awareness.
Clinical Error Recognition Performance | Baseline (T0): Prior to the educational intervention (Day 0) Post-intervention (T1): Within 1 week after completion of the intervention Follow-up (T2): During the first week of surgical clinical practice
  Change in clinical error recognition performance assessed using scenario-based clinical error recognition tests evaluating students' ability to identify patient safety risks and potential clinical errors. Outcome Measure: Total score on the Clinical Error Recognition Test, ranging from 0 to 100, where higher scores indicate better clinical error recognition performance.

SECONDARY OUTCOMES:
Clinical Decision-Making Under Stress | Baseline (T0): Prior to the educational intervention (Day 0) Post-intervention (T1): Within 1 week after completion of the intervention Follow-up (T2): During the first week of surgical clinical practice
  Change in clinical decision-making performance under stress assessed using scenario-based decision-making evaluations simulating stressful surgical clinical situations. Outcome Measure: Total score on the Clinical Decision-Making Under Stress Assessment, ranging from 0 to 100, where higher scores indicate better clinical decision-making performance under stress.
Perceived Readiness and Self-Confidence for Clinical Practice | Baseline (T0): Prior to the educational intervention (Day 0) Post-intervention (T1): Within 1 week after completion of the intervention Follow-up (T2): During the first week of surgical clinical practice
  Change in perceived readiness and self-confidence for surgical clinical practice measured using the Clinical Practice Readiness and Self-Confidence Scale. Outcome Measure: Total score on the Clinical Practice Readiness and Self-Confidence Scale, ranging from 1 to 5, where higher scores indicate greater perceived readiness and self-confidence.
Acceptability of the Digital Microlearning Program | Post-intervention (T1): Within 1 week after completion of the intervention
  Participant satisfaction and perceived usefulness of the digital microlearning program assessed using a post-intervention program acceptability questionnaire in the intervention group. Outcome Measure: Total score on the Program Acceptability Questionnaire, ranging from 1 to 5, where higher scores indicate greater acceptability and perceived usefulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Agri Ibrahim Cecen University Faculty of Health Sciences, AĞRI, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves student participants and includes questionnaire-based and educational performance data. Sharing individual-level data could pose risks to participant confidentiality and privacy. All data will be used solely for the purposes of this study and reported in aggregate form.

REFERENCES:
- [Background] World Health Organization. Patient safety curriculum guide: Multi-professional edition. Geneva: WHO; 2011.
- [Background] Lee SE, Morse BL, Kim NW. Patient safety educational interventions: A systematic review with recommendations for nurse educators. Nurs Open. 2022 Jul;9(4):1967-1979. doi: 10.1002/nop2.955. Epub 2021 May 28. PMID 34047058
- [Background] De Gagne JC, Park HK, Hall K, Woodward A, Yamane S, Kim SS. Microlearning in Health Professions Education: Scoping Review. JMIR Med Educ. 2019 Jul 23;5(2):e13997. doi: 10.2196/13997. PMID 31339105
- See also: World Health Organization resources providing background information on patient safety principles relevant to the study protocol. — https://www.who.int/teams/integrated-health-services/patient-safety